CLINICAL TRIAL: NCT02573753
Title: The Effects of Sleep on Human Microbiota: Implications for Health and Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, M.D., Ph.D., Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 15-002092
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Crossover; Single group
Oversight: Data Monitoring Committee: No

ARMS (3):
- sleep restriction (Experimental): Sleep restriction
  Interventions: Behavioral: Sleep restriction
- normal sleep (No Intervention): Normal sleep
- weight gain (Experimental): Weight gain
  Interventions: Dietary Supplement: Weight gain

INTERVENTIONS:
Behavioral: Sleep restriction
  Arms: sleep restriction
Dietary Supplement: Weight gain
  Arms: weight gain

SUMMARY:
The aggregate of microorganisms inhabiting the human body can be regarded as a dynamic reflector of both healthy and disease states, altering in response to changes in the environment. This may precede clinically detectable disease; and thereby, could be used to predict disease onset and additionally monitor response to treatment and predict prognosis. The primary hypothesis of this pilot study is that the human microbial communities are influenced by sleep and altered in humans with abnormal sleep patterns, and they may ultimately relate to disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who are eligible for ongoing IRB-approved studies will be deemed eligible for this protocol.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Subjects who are ineligible for ongoing IRB-approved studies will not be included in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2015-10; Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Changes in human microbiota induced by sleep manipulation in healthy subjects | 1 year
Changes in human microbiota induced by fluctuations in body weight and sleep in healthy subjects | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No